CLINICAL TRIAL: NCT04521049
Title: A New Clinical Utility for Tubular Markers to Identify Kidney Responders to Saxagliptin Treatment in Patients With Diabetic Nephropathy
Brief Title: Tubular Markers in Response to Saxagliptin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Marwa Mohsen Mahmoud, principal investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tubular markers
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: saxagliptin; uNGAL; u L-FABP; DKD
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- saxagliptin (Active Comparator): patients received 5 mg daily ( 2.5 mg daily dose was given to patients with an eGFR of <50 mL/min/1.73 m2
  Interventions: Drug: Saxagliptin 5mg
- control (No Intervention): patients received the antihyperglycemic medication(s) such as metformin and/or sulphonyl ureas or insulin with no added gliptins,

INTERVENTIONS:
Drug: Saxagliptin 5mg — Patients would be assigned to saxagliptin (Onglyza® AstraZeneca Pharmaceuticals LP, Indiana, USA), either received a dose of 5 mg or 2.5 mg daily if patients had eGFR <50 mL/min/1.73 m2
  Other Names: Onglyza
  Arms: saxagliptin

SUMMARY:
the study aims to investigate whether treatment with saxagliptin would induce beneficial changes in renal NGAL and L-FABP biomarkers and if they would be used as a tool to identify patients' categories with a particular renal response to DPP-4inhibition. Secondly, to find an association between NGAL and L-FABP, and the relevant renal parameters for both baseline values and rate of changes across defined time points.

DETAILED DESCRIPTION:
Diabetic kidney disease (DKD) is considered a substantial cause of end-stage kidney disease (ESKD) worldwide. Incorporation of renoprotective options during interventions to prevent the development of DKD and attenuation of its progression; is of the utmost importance. Incretin-based therapies, specifically dipeptidyl peptidase 4 (DPP-4) inhibitors exhibited albuminuria lowering potential beyond their antihyperglycemic effects. Saxagliptin, a potent selective DPP-4 inhibitor which has been used as monotherapy or in combination with antidiabetics, has demonstrated great renal efficiency on both experimental and clinical scale .

Although albumin excretion rate (AER) is a powerful predictor of kidney function deterioration and progressive renal dysfunction, it is primarily a marker of glomerular damage and it has some drawbacks. For example; some patients may follow a non-albuminuric pathway to kidney impairment, others do not progress to macroalbuminuria but remain at microalbuminuria or even regress to normoalbuminuria. Thus, more sensitive and specific renal biomarkers than AER will be valuable in predicting early kidney injury and the progression of diabetic renal damage.

Besides glomerular damage, tubulointerstitial dysfunction largely contributes to the pathology of diabetic nephropathy. Neutrophil gelatinase-associated lipocalin (NGAL) and liver type fatty acid binding protein (L-FABP) are apparent as excellent biomarkers of tubular damage and are earlier predictors of acute kidney injury relative to microalbuminuria. NGAL is produced by neutrophils, highly expressed in tubular epithelium and released from tubular cells following damage . L-FABP is expressed in the proximal tubules and secreted into urine upon tubulointerstitial damage. Clinical significance of these biomarkers lies in their emergence in normoalbuminuric patients and their association with increased albuminuria and progression to ESRD with sustained high urinary markers' levels.

ELIGIBILITY:
Inclusion Criteria:

* T2 DM,
* prevalent albuminuria (30-3000mg/g),
* controlled hypertension (defined as blood pressure <140/90 mm Hg) on a selected angiotensin receptor blocker, olmesartan 20mg/day for at least 4 weeks before intervention.

Exclusion Criteria:

* type 1 diabetes,
* poorly controlled hypertension (140-160/90-100 mm Hg),
* pancreatitis,
* malignancies
* albuminuria more than 3000mg/g.
* cardiovascular diseases (acute myocardial infarction, cerebrovascular disease in the past 6months,
* End Stage Renal Disease (ESRD) on chronic dialysis, renal transplant, a serum creatinine >6.0 mg/dL, or estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
to measure renal effect of saxagliptin on tubular markers | 3 months
  the rate of change of uNGAL and u LFABP markers would be estimated across the two time points after saxagliptin treatment .
to measure effect of saxagliptin on renal on albuminuria | 3 months
  the rate of change of UACR would be measured across the two time points after saxagliptin treatment
to classify renal responders to saxagliptin using tubular markers | 3 months
  patients would be classified into high risk and low risk patients according to their marker levels

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Elberry, prof, Study Chair — Clinical Pharmacology Faculty of Medicine, Beni-Suef University, Beni-Suef, Egypt
Locations (1):
- Faculty of Pharmacy, Al Qāhirah al Jadīdah, Egypt

REFERENCES:
- See also: Urinary Proteomics as a Tool to Identify Kidney Responders to Dipeptidyl Peptidase-4 Inhibition: A Hypothesis-Generating Analysis from the MARLINA-T2D Trial — http://onlinelibrary.wiley.com/doi/full/10.1002/prca.201800144